CLINICAL TRIAL: NCT03687840
Title: Evaluation of Spatio-Temporal Gait Parameters and Gait Symmetry In Diabetic Polyneuropathic Individuals With Lower Extremity Burn Injury
Brief Title: Spatio-Temporal Gait Parameters and Gait Symmetry In Diabetic Lower Extremity Burn Injury.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other); Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Melek Merve ERDEM, Research Assistant, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GO 17/07
Record Dates: First submitted 2018-08-22; First posted 2018-09-27 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Polyneuropathy; Foot Injuries
Keywords: Diabetic Polyneuropathy; Lower Extremity Burn Injury; Spatio-Temporal Parameters of Gait; Gait Symmetry
MeSH Terms: conditions — Diabetic Neuropathies; Foot Injuries | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Other): Spatio-Temporal gait analysis of subjects with unilateral lower extremity burn injuries due to diabetic polyneuropathy.
  Interventions: Diagnostic Test: gait analysis
- Control Group (Other): Spatio-Temporal gait analysis of subjects with only diabetic polyneuropathy.
  Interventions: Diagnostic Test: gait analysis

INTERVENTIONS:
Diagnostic Test: gait analysis — Computerized gait analysis system was used to 3 times to evaluate the spatio-temporal parameters of gait.

SUMMARY:
This study evaluated the spatio-temporal gait parameters and gait symmetry in individuals with lower extremity burn injury due to diabetic polyneuropathy. Study group consisted of 14 subjects with unilateral lower extremity burn injuries due to diabetic polyneuropathy and control group consisted of 14 subjects with only diabetic polyneuropathy.

DETAILED DESCRIPTION:
Diabetic polyneuropathy, a frequent complication of diabetes, is used to describe sensory, motor and autonomic nerve damage caused by metabolic and micro vessel alterations due to hyperglycaemia. The signs and symptoms of diabetic polyneuropathy vary according to the type of nerve fiber affected. The involvement of the small nerve fibers results in deterioration of the pain and temperature perception, while the impairing of large nerve fibers result in decrease of touch and proprioception sensations. Due to the sensory loss, accidental foot injuries may develop in patients with diabetic polyneuropathy. While the feet constitute a small percentage (3.5%) of the total body surface area, burn injuries of them in patients with diabetic polyneuropathy can cause significant effects on quality of life because impaired wound healing process in diabetics may cause risk of prolonged bed rest and hospitalization period, and increased early and late complications. Therefore, it has an important effects on daily living activities because it causes inadequacies in gait and balance activities due to the negative effects on mobility and weight bearing functions. In studies that examining changes in gait parameters in other diabetic foot complications such as sensory loss, ulceration, and amputation as secondary to diabetic polyneuropathy have shown that these individuals acquire a protective adaptive gait strategies that allow for more controlled gait in the present of proprioceptive deficits such as slower gait speed, smaller step length and in particular increased opposite foot off time in order to shift body weight from injured limb to unaffected side. There's no studies have yet been conducted to investigating of changes in gait parameters in patients who have diabetic polyneuropathy-related lower extremity burn injury. The aim of this case-control study is to examine whether similar gait strategies have been gained in this group of patients, as indicated in the results of previous studies demonstrating protective adaptive gait strategies that adopt under the presence of other diabetic foot complications due to diabetic polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Study group, include cases with a diagnosis of diabetic polyneuropathy and unilateral lower limb burn injury.
* Control group consists of adults with a confirmed diagnosis of diabetic polyneuropathy without burn injury.

Exclusion Criteria:

* presence of active ulcerations
* presence of other diabetic morbidities (nephropathy, retinopathy, vestibulopathy)
* orthopedic, musculoskeletal, neurological problems or previous surgical interventions that may affect the mobility and original gait dynamics except for diabetic polyneuropathy,
* using of assistive devices
* body mass index> 40 kg/m²

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-02-11 (Actual); Study Completion 2018-03-11 (Actual)

PRIMARY OUTCOMES:
Step Length | 1 week
  It is measured along the length of the walkway, from the heel center of the current footprint to the heel center of the previous footprint on the opposite foot.The unit of measure is centimeters.

SECONDARY OUTCOMES:
Stride Length | 1 week
  It is measured on the line of progression between the heel points of two consecutive footprints of the same foot (left to left, right to right). The unit of measure is centimeters.
Step Width | 1 week
  It is measured from the midline midpoint of the current footprint to the midline midpoint of the previous footprint on the opposite foot.The unit of measure is centimeters.
Foot Progression Angle | 1 week
  It is the angle between the line of progression and the midline of the footprint. This angle is zero if the geometric mid- line of the footprint is parallel to the line of progression; positive, toe-out, when the mid-line of the footprint is outside the line of progression and negative, toe-in, when inside the line of progression. The unit of measure is degrees.
Speed | 1 week
  It is obtained after dividing the distance traveled by the ambulation time. It is expressed in centimeters per second (cm/sec)
Cadence | 1 week
  The rate at which a person walk, expressed in steps per minute (step/min). The average cadence is 100 - 115 steps/min.
Percentage of Double Support | 1 week
  It is the amount of time that a person spends with both feet on the ground during one gait cycle. It is presented as a percentage of the gait cycle time (% gait cycle). The percentage of time spent in double support decreases as the speed of walking increases.
Percentage of Stance | 1 week
  The stance phase is the weight bearing portion of each gait cycle. It is initiated by heel contact and ends with toe off of the same foot. It is the time elapsed between the first contact and the last contact of two consecutive footfalls on the same foot. It is also presented as a percentage of the gait cycle time (% gait cycle)
Percentage of Swing | 1 week
  It is initiated with toe off and ends with heel strike. It is the time elapsed between the last contact of the current footfall to the first contact of the next footfall on the same foot. It is expressed in seconds (sec) and it is also presented as a percent of the gait cycle (% gait cycle) of the same foot. The Swing Time is equal to the Single Support time of the opposite foot.
Symmetry Index | 1 week
  It's calculated in order to evaluate symmetry and bilateral coordination of gait. The Symmetry Index and Symmetry Angle are interpreted as a complete symmetry if the result is 0. Evaluation of asymmetries observed in the spatio-temporal characteristics, a deviation of at least 10% from the 0 value for exact symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Melek M. ERDEM, PT, M.Sc., Principal Investigator — Tayyip Erdogan University Training and Research Hospital; Semra TOPUZ, Assoc. Prof., Study Director — Hacettepe University; Kemal KISMET, Assoc. Prof., Study Director — Ankara Training and Research Hospital; Gonul KOC, MD, Study Chair — Ankara Training and Research Hospital; Ahmet C. YASTI, Prof., Study Chair — Numune Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Training and Research Hospital, Ankara, Cankaya
  - Numune Training and Research Hospital, Ankara, Cankaya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within 6 months with completion of the result report.
Access Criteria: Requestors will be required to sign a Data Access Agreement.
URL: https://www.researchgate.net/profile/Melek_Erdem2

REFERENCES:
- [Background] Jones LM, Coffey R, Khandelwal S, Atway S, Gordillo G, Murphy C, Fries JA, Dungan K. A clinician's guide to the treatment of foot burns occurring in diabetic patients. Burns. 2014 Dec;40(8):1696-701. doi: 10.1016/j.burns.2014.01.026. Epub 2014 Mar 20. PMID 24656951